CLINICAL TRIAL: NCT00875225
Title: Culturally Sensitive Intervention: CSI Birmingham
Brief Title: Using Multimedia Technology for Hypertension Control for Low-Income African Americans
Acronym: CSI Birmingham
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cooper Green Mercy Hospital (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sandral Hullett, MD/Medical Director, Cooper Green Mercy Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 59741 - Finding Answers
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2009-04

CONDITIONS: Hypertension
Keywords: Hypertension; Adherence to medications
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control DVD (Active Comparator): Control DVD with usual care information
  Interventions: Behavioral: DVD
- Intervention DVD (Active Comparator): Intervention group will receive DVD with patient stories and information from health care professionals
  Interventions: Behavioral: Intervention DVD

INTERVENTIONS:
Behavioral: DVD — Control group will receive usual care DVD from health professionals
  Arms: Control DVD
Behavioral: Intervention DVD — Intervention group will receive intervention DVD with patient stories and information from health care professionals
  Arms: Intervention DVD

SUMMARY:
The purpose of this study is to test an interactive DVD intervention to encourage patients to stick to their blood pressure medication in order to achieve blood pressure control for African American patients. The intervention will convey health messages through personal patient stories who have dealt with or continue to struggle with high blood pressure.

Hypothesis 1: At the end of 9 months a higher proportion of patients randomized to the intervention group will achieve appropriate blood pressure control.

Hypothesis 2: At the end of 9 months a higher proportion of patients who randomized to the intervention group will report high adherence to their hypertension medications.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Clinical Diagnosis of Hypertension
* Patient at Cooper Green Hospital
* Provided Informed Consent
* Age 18 or older

Exclusion Criteria:

* Pregnant
* Diagnosed with dementia, schizophrenia, bipolar illness, or other serious acute or chronic medical co-morbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2006-12; Primary Completion 2009-05 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Blood pressure control | Two years

SECONDARY OUTCOMES:
Adherence to hypertension medications | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Sandral Hullett, MD, Principal Investigator — Cooper Green Mercy Hospital
Locations (1):
- Cooper Green Mercy Hospital, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Houston TK, Allison JJ, Sussman M, Horn W, Holt CL, Trobaugh J, Salas M, Pisu M, Cuffee YL, Larkin D, Person SD, Barton B, Kiefe CI, Hullett S. Culturally appropriate storytelling to improve blood pressure: a randomized trial. Ann Intern Med. 2011 Jan 18;154(2):77-84. doi: 10.7326/0003-4819-154-2-201101180-00004. PMID 21242364